CLINICAL TRIAL: NCT00032058
Title: MR Imaging And MR Spectroscopic Imaging Of Prostate Cancer Prior To Radical Prostatectomy: A Prospective Multi-Institutional Clinicopathological Study
Brief Title: Magnetic Resonance Imaging and Magnetic Resonance Spectroscopic Imaging in Diagnosing the Extent of Disease in Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000069254; ACRIN-6659
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2005-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: magnetic resonance imaging
Procedure: magnetic resonance spectroscopic imaging

SUMMARY:
RATIONALE: Imaging procedures such as magnetic resonance imaging (MRI) and magnetic resonance spectroscopic imaging (MRSI) may improve the ability to detect the extent of prostate cancer. It is not yet known if MRI combined with MRSI is more effective than MRI alone in detecting the extent of prostate cancer.

PURPOSE: Diagnostic trial to compare the effectiveness of combining MRI with MRSI to that of MRI alone in determining the extent of prostate cancer in patients who are scheduled to undergo surgery to remove the prostate gland.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the accuracy of MRI vs MRI combined with magnetic resonance spectroscopic imaging (MRSI) for the localization of prostate cancer prior to radical prostatectomy in patients with stage I or II adenocarcinoma of the prostate.
* Compare the incremental benefit of these tests on diagnostic accuracy in these patients.
* Compare the incremental benefit of MRSI for interobserver agreement vs MRI alone in the localization of prostate cancer in these patients.
* Compare the accuracy of combined MRSI with that of other available information on tumor extent derived from digital rectal exam, PSA level, Gleason score, and Partin nomogram in these patients.

OUTLINE: This is a multicenter study.

At least 6 weeks after biopsy, patients undergo MRI and magnetic resonance spectroscopic imaging (MRSI) over approximately 1 hour. Within 6 months of MRI/MRSI, patients undergo radical prostatectomy.

PROJECTED ACCRUAL: A total of 134 patients will be accrued for this study within 7 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage I-II adenocarcinoma of the prostate

  * At least 6 weeks since prior biopsy
* Scheduled to undergo radical prostatectomy within 6 months of MRI and magnetic resonance spectroscopic imaging (MRSI)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No cardiac pacemakers

Other:

* Must be willing and able to undergo MRI/MRSI
* No allergy to latex
* No contraindications to MRI such as non-compatible intracranial vascular clips
* No metallic hip implant or any other metallic implant or device that would compromise quality of MRI/MRSI
* No contraindications to or intolerance of endorectal coil insertion (e.g., prior abdominoperineal resection of the rectum or Crohn's disease)
* No general medical or psychiatric condition or physiologic status unrelated to prostate cancer that would preclude valid informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior BCG for bladder cancer

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior androgen-deprivation therapy

Radiotherapy:

* No prior prostatic or rectal radiotherapy

Surgery:

* See Disease Characteristics
* No prior cryosurgery
* No prior surgery for prostate cancer
* No prior transurethral resection of the prostate (TURP)
* No prior rectal surgery

Other:

* No prior complementary alternative medicine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weinreb, MD, Study Chair — Yale University
Locations (8):
- United States (8):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas